CLINICAL TRIAL: NCT00006457
Title: Clinical Phase I Multiple-Dose Safety Research Study of Oltipraz in Smokers
Brief Title: Oltipraz in the Prevention of Lung Cancer in People Who Smoke
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Masking: Double | Purpose: Prevention
Other Study IDs: NCI 00L1; NU-00L1; DUMC-000346-00-2; NCI-P00-0167
Record Dates: First submitted 2000-11-06; First posted 2003-05-30 (Estimated); Last update posted 2012-06-11 (Estimated); Status verified 2012-06

CONDITIONS: Lung Cancer
Keywords: non-small cell lung cancer; small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung; Small Cell Lung Carcinoma | interventions — oltipraz

INTERVENTIONS:
Drug: oltipraz

SUMMARY:
RATIONALE: Chemoprevention therapy is the use of certain drugs to try to prevent the development of cancer.

PURPOSE: Randomized phase I trial to study the effectiveness of oltipraz in preventing lung cancer in people who smoke.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the effect of oltipraz on the level of BP-7,8-diol-9,10-epoxide (BPDE) DNA adducts in the lung lining cells (macrophages and bronchial epithelial cells) of smokers.
* Determine the tolerability and toxicity of this treatment regimen in these patients.
* Determine the effect of this treatment regimen on the level of macromolecule adducts in the blood (e.g., BPDE DNA, BPDE hemoglobin, and 8-hydroxy-deoxyguanine), oral lining cells (BPDE DNA), bladder lining cells (4-aminobiphenyl DNA), and lung macrophages (8-hydroxy-deoxyguanine) in these patients.
* Determine the effect of this treatment regimen on the change (decrease) in activation of NNK as measured by change (increase) in urinary NNAL plus NNAL glucuronide in these patients.
* Determine the effect of this treatment regimen on the oxidative state, glutathione-S-transferase activity, and superoxide dismutase 3 and phase II enzymes in the lungs and blood of these patients.
* Compare the changes in oxidative state and phase II enzymes with changes in adduct levels in the lungs and blood of these patients.
* Determine the correlation between oltipraz-induced changes in phase II enzymes and adduct formation with genotypic variation in glutathione-S-transferase isozymes in these patients.
* Compare the response to this treatment regimen in terms of oxidative state, phase II enzymes, and adduct formation in the lungs vs the blood in these patients.

OUTLINE: This is a randomized, double-blind, multicenter study. Patients are stratified according to participating center. Patients are randomized to one of three treatment arms.

* Arm I: Patients receive an oral placebo weekly.
* Arm II: Patients receive low-dose oral oltipraz weekly.
* Arm III: Patients receive high-dose oral oltipraz weekly. Treatment continues for 12 weeks in the absence of unacceptable toxicity.

Patients are followed at 4 weeks.

PROJECTED ACCRUAL: A total of 66 patients (22 per treatment arm) will be accrued for this study within 21 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Current cigarette smokers

  * At least 20 cigarettes a day
  * No variation of more than 10 in the number of cigarettes smoked per day within the past 3 months
  * At least 10 years of smoking any amount
  * Failed to stop smoking after at least one attempt to quit within the last 3 years
* Prior stage I non-small cell lung cancer allowed if surgically resected with at least a lobectomy
* No concurrent evidence of lung cancer
* Willing to undergo 2 bronchoscopies

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* ECOG 0

Life expectancy:

* Not specified

Hematopoietic:

* CBC normal
* Hemostasis normal

Hepatic:

* PT and PTT normal

Renal:

* Blood chemistries normal
* Nonfasting glucose no greater than 200 mg/dL
* No active renal disease
* No urinary tract infection by urinalysis (trace protein allowed)

Cardiovascular:

* EKG normal
* No coronary artery disease requiring continuous medication

Pulmonary:

* Chest radiograph normal (postsurgical changes allowed)
* No acute or significant chronic abnormality
* FEV1 greater than 1.8 L or 75% predicted
* No chronic obstructive pulmonary disease requiring continuous medication

Other:

* No known hypersensitivity or prior adverse reaction to oltipraz
* No inmates or prisoners
* No medical or psychological condition that would preclude study (e.g., acute psychosis)
* No prior malignancy except nonmelanomatous skin cancer, cervical dysplasia, or curatively treated stage I or II cancer of the head and neck
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 6 months after study

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* At least 3 months since prior potential chemoprevention agent (e.g., oltipraz, retinoids, or acetylcysteine)

Endocrine therapy:

* Not specified

Radiotherapy:

* Not specified

Surgery:

* See Disease Characteristics

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2000-08; Primary Completion 2004-04 (Actual); Study Completion 2004-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Raymond C. Bergan, MD, Study Chair — Robert H. Lurie Cancer Center
Locations (2):
- United States (2):
  - Robert H. Lurie Comprehensive Cancer Center, Northwestern University, Chicago, Illinois
  - Duke Comprehensive Cancer Center, Durham, North Carolina